CLINICAL TRIAL: NCT06298591
Title: The Efficacy of Subcision in Combination With PRP Injection and Fractional Co2 Laser in Treatment of Atrophic Scar: Clinical and Ultrasonic Study
Brief Title: The Efficacy of Combination Therapy in Atrophic Scars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Ahmed Hasan, Assistant Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: atrophic scar treatment
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Atrophic Scar
MeSH Terms: interventions — Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subcision (Other)
  Interventions: Procedure: co2 laser

INTERVENTIONS:
Procedure: co2 laser — laser
  Other Names: fractional co2 laser

SUMMARY:
There are more than 100 million patients who develop scar formation caused by various factors, such as post-inflammatory acne and trauma (1). They often have physical, aesthetic, psychological, and social barriers. Scar tissue is naturally a stage of wound healing. Abnormal wound healing produces a spectrum of scar tissue types such as atrophic, hypertrophic, and keloid scars (2).

Atrophic scars are dermal depressions, which are commonly caused by the destruction of collagen following inflammatory process. This permanent disfiguring sequelae correlates with the duration of pathology, severity of lesion, and delay in therapy (3).

Treatment of atrophic acne scars remains a therapeutic challenge, yet there is no standard option as the most effective treatment (4). A range of possible options has been investigated including surgical techniques (subcision, non-ablative laser treatment, resurfacing techniques (ablative laser treatment, dermabrasion), and injection or dermal fillers or fat, and a combination of two or more modalities (5).

Ultrasound is a unique non-invasive and non-radiating medical imaging tool in the investigation of dermatological diseases by providing detailed anatomic and physiologic data of skin lesions and deeper soft tissue changes. Lesion size in three dimensions-lengths, width, and depth, morphology, the detailed anatomic information provided by sonography is useful to assessment of effect of different types of treatment modality to improve atrophic scar and avoid invasive assessment tools as punch biopsy for histopathological examination (6)

DETAILED DESCRIPTION:
atrophic scar mangment

ELIGIBILITY:
Inclusion Criteria:

- Patients aged from 12 to 60 years with

* post inflammatory atrophic scar.
* post traumatic atrophic scar.
* post operative atrophic scar

Exclusion Criteria:

* post acne scar.
* active skin infection.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
change of dermal thickness in sonar and Vancouver scale | 3 years
  objective